CLINICAL TRIAL: NCT00012298
Title: Phase I/II Study of Two Sequential Doses of IDEC-Y2B8 in Patients With Relapsed Low-Grade and Follicular Non-Hodgkin's Lymphoma
Brief Title: Radiolabeled Monoclonal Antibody Plus Rituximab With and Without Filgrastim and Interleukin-11 in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial completed prematurely.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00008; NCI-2009-00008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068503; MC998C (Other: Mayo Clinic); 312 (Other: CTEP); NCT01646879 (obsolete NCT alias)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; ibritumomab tiuxetan; Indium; oprelvekin; Interleukin-11; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (radiolabeled monoclonal antibody therapy) (Experimental): Patients receive rituximab IV on days 1 and 8, indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1, and yttrium Y 90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8. Patients also receive filgrastim (G-CSF) subcutaneously (SC) and interleukin-11 SC until blood counts recover.
  Interventions: Biological: rituximab; Biological: yttrium Y 90 ibritumomab tiuxetan; Biological: indium In 111 ibritumomab tiuxetan; Biological: oprelvekin; Biological: filgrastim

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Biological: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan
Biological: indium In 111 ibritumomab tiuxetan — Given IV
  Other Names: IDEC-In2B8
Biological: oprelvekin — Given subcutaneously
  Other Names: adipogenesis inhibitory factor; IL-11; interleukin 11; Neumega
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen

SUMMARY:
Phase I/II trial to study the effectiveness of combining radiolabeled monoclonal antibody therapy and rituximab with and without filgrastim and interleukin-11 in treating patients who have relapsed or refractory non-Hodgkin's lymphoma. Radiolabeled monoclonal antibodies can locate cancer cells and deliver cancer-killing substances to them without harming normal cells. Biological therapies such as filgrastim and interleukin-11 use different ways to stimulate the immune system and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of yttrium Y 90 ibritumomab tiuxetan (IDEC-90Y2B8) administered with rituximab with and without filgrastim (G-CSF) and interleukin-11 (IL-11) in patients with relapsed low-grade or follicular CD20+ non-Hodgkin's lymphoma. (Phase I) II. Determine the toxicity of this regimen in these patients. III. Determine the response rate in patients treated with this regimen. IV. Compare tumor and normal organ dosimetry with positron emission tomography and computerized tomography scans, subsequent tumor response, and normal organ toxicity by utilizing indium In 111 ibritumomab tiuxetan radioimmunoconjugate scans before each IDEC-90Y2B8 dose in these patients. (Phase I) V. Determine the immune response to this regimen, in terms of human anti-mouse and human anti-chimeric antibody formation, in these patients. (Phase I) VI. Determine whether G-CSF and IL-11 can ameliorate the effect of the MTD of IDEC-90Y2B8 on bone marrow function in these patients. (Phase I) VII. Determine progression-free survival at 3 years. (Phase II)

OUTLINE:

PHASE I: Patients receive rituximab IV on days 1 and 8, indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1 (for radioimaging), and IDEC-90Y2B8 IV over 10 minutes on day 8. Treatment repeats 24-36 weeks later for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Once the maximum tolerated dose (MTD) of IDEC-90Y2B8 is determined, patients also receive filgrastim (G-CSF) subcutaneously (SC) daily beginning when absolute neutrophil count is less than 1,500/mm3 and continuing until blood counts recover. Patients also receive interleukin-11 (IL-11) SC beginning when platelet count is less than 75,000/mm^3 and continuing until blood counts recover. Patients undergo PBSC transplantation only if marrow recovery is inadequate.

Cohorts of 3-6 patients receive escalating doses of IDEC-90Y2B8 until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to determine the MTD of this radioimmunotherapy with the addition of the prophylactic cytokines, G-CSF and IL-11.

PHASE II: Patients receive rituximab, indium In 111 ibritumomab tiuxetan, and IDEC-90Y2B8 IV as determined at the MTD in phase I. Treatment repeats 24-36 weeks later for a total of 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven relapsed or refractory low-grade or follicular CD+ non-Hodgkin lymphoma, including 1 of the following:

  * Small lymphocytic lymphoma
  * Lymphoplasmacytoid lymphoma
  * Follicular center lymphoma (grades I, II, and III)
  * Extranodal marginal zone B-cell lymphoma
  * Nodal marginal zone B-cell lymphoma
  * Splenic marginal zone B-cell lymphoma (monocytoid B-cell lymphoma)
* Less than 25% bone marrow involvement of cellular marrow with lymphoma by bilateral bone marrow aspirate and biopsy
* ECOG performance status 0-2
* Bidimensionally measurable disease with at least 1 lesion >= 2 cm in the greatest diameter
* No prior myeloablative therapy with autologous or allogeneic bone marrow transplantation or peripheral blood stem cell support
* No concurrent corticosteroid therapy, except prednisone (or equivalent) for adrenal failure or < 20mg of prednisone daily
* No prior external beam radiotherapy to >25% of active bone marrow
* More than 4 weeks since prior surgery other than diagnostic surgery
* No other concurrent myelosuppressive antineoplastic agents
* No prior radioimmunotherapy, including yttrium Y 90 ibritumomab tiuxetan or iodine I 131 monoclonal antibody tositumomab or Lym-1
* No CNS lymphoma
* No myelodysplastic syndromes or marrow chromosomal changes suggesting myelodysplasia
* No HIV or AIDS-related lymphoma
* No pleural effusion or ascites with lymphoma cells
* No active infection
* No other serious non-malignant disease that would preclude study participation
* No other active primary malignancy
* No known human anti-mouse or human anti-chimeric antibody
* No prior skin rash (e.g., Stevens-Johnsons syndrome or toxic epidermal necrolysis) from rituximab therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 150,000/mm^3
* Total lymphocyte count < 5,000/mm^3 for patients with small lymphocytic lymphoma
* Bilirubin =< 2 mg/dL
* Creatinine =< 2 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2001-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Witzig, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I is a series of three single-arm trials: Trial 1 will determine the Y2B8 MTD without growth factors, Trial 2 will test the regimen with G-CSF and IL-11 added to the treatment, and Trial 3 tests different levels of IL-11 in the regimen.
Groups:
- Treatment: Trial 1, Dose Level 1: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.2 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
- Treatment: Trial 1, Dose Level 2: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
- Treatment: Trial 2, Dose Level 3: Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.2 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 75,000.
- Treatment: Trial 2, Dose Level 4: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 75,000.
- Treatment: Trial 3, Dose Level 5: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Cycle 2 (Cycle 2 delivered 24-36 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 150,000.
- Treatment: Trial 3, Dose Level 6; Treatment : Phase II (Dose Level 6): Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Cycle 2 (Cycle 2 delivered 24-36 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 150,000.
Period: Overall Study
Arm/Group | Treatment: Trial 1, Dose Level 1 | Treatment: Trial 1, Dose Level 2 | Treatment: Trial 2, Dose Level 3 | Treatment: Trial 2, Dose Level 4 | Treatment: Trial 3, Dose Level 5 | Treatment: Trial 3, Dose Level 6 | Treatment : Phase II (Dose Level 6)
Started | 11 | 7 | 9 | 4 | 5 | 6 | 39
Completed | 11 | 7 | 9 | 4 | 5 | 6 | 39
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Trial 1, Dose Level 1: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.2 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
- Treatment: Trial 1, Dose Level 2: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
- Treatment: Trial 2, Dose Level 3: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.2 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 75,000.
- Treatment: Trial 2, Dose Level 4: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 75,000.
- Treatment: Trial 3, Dose Level 5: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 24-36 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 150,000.
- Treatment: Trial 3, Dose Level 6; Treatment : Phase II (Dose Level 6): Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 24-36 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 150,000.
- Total: Total of all reporting groups
Arm/Group | Treatment: Trial 1, Dose Level 1 | Treatment: Trial 1, Dose Level 2 | Treatment: Trial 2, Dose Level 3 | Treatment: Trial 2, Dose Level 4 | Treatment: Trial 3, Dose Level 5 | Treatment: Trial 3, Dose Level 6 | Treatment : Phase II (Dose Level 6) | Total
Number analyzed (Participants) | 11 | 7 | 9 | 4 | 5 | 6 | 39 | 81
Age, Continuous [Median (Full Range); unit: years] | 60 [39 to 70] | 56 [31 to 65] | 52 [37 to 70] | 51 [30 to 67] | 46 [42 to 60] | 59 [28 to 62] | 58 [36 to 76] | 58 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 2 | 3 | 1 | 17 | 33
  Male | 7 | 3 | 7 | 2 | 2 | 5 | 22 | 48
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Croatia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  United States | 10 | 7 | 9 | 3 | 5 | 6 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Yttrium Y-90 Ibritumomab Tiuxetan (Y2B8) With and Without Filgrastim (G-CSF) and Interleukin-11 (IL-11) (Phase I)
Description: This study is a series of 3 single-arm phase-I trials designed to determine the maximum tolerated dose (MTD) of a 2-cycle combination regimen containing Rituxan + Y2B8 radioimmunotherapy with and without the use of G-CSF and IL-11. Trial 1 will determine the Y2B8 MTD in the combined regimen without growth factors. Trial 2 will evaluate the combined regimen with growth factors. Trial 3 starts IL-11 earlier (when platelet count drops below 150000) and reduces the dosing interval to twice weekly.
  > Dose-limiting toxicity (DLT) is defined as an adverse event in the second cycle attributed to treatment and meeting the following criteria: Grade 4 ANC or platelet decrease for 14 days, or grade 3 for 28 days, or any other grade 3 Non-Heme event.
  > If at any time 2 or more patients (of a maximum of 6) at any dose level experience DLT, then the MTD will be defined as the previous dose level during that trial. The number of patients with a DLT are reported here.
Time Frame: At 8 weeks
Population: DLTs were determined in the second cycle of combined treatment. Only Phase I patients that were evaluated after 2 cycles of treatment are included in this evaluation. Two patients at Dose Level 1, 1 patient at Dose Level 2, 4 patients at Dose Level 3, and 1 patient at Dose Level 5 were not evaluated for MTD.
Measure: Number; unit: Patients reporting Dose-Limiting Events
Groups:
- Treatment: Trial 2, Dose Level 3: Patients receive:
  Cycle 1:
  50 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 12-24 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.2 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 75,000.
Arm/Group | Treatment: Trial 1, Dose Level 1 | Treatment: Trial 1, Dose Level 2 | Treatment: Trial 2, Dose Level 3 | Treatment: Trial 2, Dose Level 4 | Treatment: Trial 3, Dose Level 5 | Treatment: Trial 3, Dose Level 6
Number analyzed (Participants) | 9 | 6 | 5 | 4 | 4 | 6
Patients reporting Dose-Limiting Events | 0 | 2 | 0 | 2 | 0 | 1

2. Primary Outcome: Toxicity of Single-dose Y2B8 Radioimmunotherapy With and Without the Use of Growth Factors (Phase I)
Description: Evaluated using the Common Toxicity Criteria (CTC) version 2.0. This data is presented as the number of patients reporting grade 3 or higher, grade 4 or higher, or grade 5 adverse events regardless of event attribution.
Time Frame: Assessed up to week 24
Population: All patients that were evaluated for adverse events after at least one cycle of treatment were used in this analysis.
Measure: Number; unit: participants
Arm/Group | Treatment: Trial 1, Dose Level 1 | Treatment: Trial 1, Dose Level 2 | Treatment: Trial 2, Dose Level 3 | Treatment: Trial 2, Dose Level 4 | Treatment: Trial 3, Dose Level 5 | Treatment: Trial 3, Dose Level 6
Number analyzed (Participants) | 11 | 7 | 9 | 4 | 5 | 6
participants
  Grade 3+ Adverse Event | 9 | 6 | 8 | 4 | 5 | 6
  Grade 4+ Adverse Event | 2 | 5 | 2 | 2 | 1 | 1
  Grade 5 Adverse Event | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Proportion of Patients Who Receive 2 Sequential Doses of Y2B8 Immunotherapy and Are Progression-free (Phase II)
Description: Estimated by the number of successes divided by the total number of evaluable patients. Exact binomial confidence intervals for the true success proportion will be calculated.
Time Frame: At 3 years
Population: Forty-five patients were registered to Dose Level 6 (39 patients registered to the Phase II portion and 6 patients registered to Dose Level 6 in the Phase I portion). Of the 45 patients, 33 patients received 2 sequential doses of Y2B8 and were evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Treatment : Dose Level 6: Patients receive:
  Cycle 1:
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
  Cycle 2 (Cycle 2 delivered 24-36 weeks after Cycle 1):
  250 mg/m^2 rituximab IV on days 1 and 8, 2 mg (5.0mCi of In-111) Indium (In-111 ibritumomab tiuxetan) IV over 10 minutes on day 1, 0.4 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8.
  Patients also receive:
  480 mcg filgrastim (G-CSF) subcutaneously (SC) daily when ANC is less than 1500.
  50 micrograms/kg Interleukin-11 SC when PLT counts less than 150,000.
Arm/Group | Treatment : Dose Level 6
Number analyzed (Participants) | 33
proportion of participants | .45 [.28 to .64]

4. Secondary Outcome: Association Between the Amounts of Tumor Radiation Indicated by the In2B8 Scan and Tumor Response (Phase I)
Description: Assessed using a correlated logistic regression model and generalized estimating equations (GEE). Covariates such as dose level and use of prophylactic cytokines may also be included in this model. A Wilcoxon test will be used to assess the equality of the distributions of the continuous levels of predicted tumor radiation from the In2B8 scans by response.
Time Frame: At week 12
Population: Not collected. Study team decision not to analyze this endpoint.
Arm/Group | Treatment (Radiolabeled Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Association Between In2B8 Scan and Positron Emission Tomography Scan Results (Phase I)
Description: Explored using a contingency table and sensitivity and specificity will be calculated using 90% exact confidence intervals.
Time Frame: At week 12
Population: Not collected. Study team decision not to analyze this endpoint.
Arm/Group | Treatment (Radiolabeled Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Appearance of Tumor and Normal Organ Images on the Second In2B8 Scan (Phase I)
Description: Calculated from the serial gamma camera images. Compared using a signed-rank-test. Scatter plots will be used to further explore relationships between these residence times and Bland- Altman methods can be used to assess the agreement between the first and second In2B8 scan residence times.
Time Frame: At week 12
Population: Not collected. Study team decision not to analyze this endpoint.
Arm/Group | Treatment (Radiolabeled Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Survival (Phase II)
Description: Estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 5 years
Population: Phase II portion of the study. One patient out of the 39 was deemed ineligible and was not included in survival analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Treatment : Dose Level 6
Number analyzed (Participants) | 38
years | NA [8.1 to NA] — Median and upper 95% confidence interval were not reached.

8. Secondary Outcome: Time to Disease Progression (Phase II)
Description: Estimated using the method of Kaplan-Meier.
Time Frame: From registration to the earliest date documentation of>disease progression, assessed up to 5 years
Population: All eligible phase II patients. One out of the 39 phase II patients was deemed ineligible.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Treatment : Dose Level 6
Number analyzed (Participants) | 38
years | 2 [1.6 to NA] — Upper 95% confidence interval was not reached.

9. Secondary Outcome: Tumor Response Rate (Phase II)
Description: Calculated by the number of tumor responses divided by the total number of evaluable patients. An exact binomial confidence interval will be calculated.
Time Frame: Assessed up to 5 years
Population: All eligible phase II patients. One of the 39 phase II patients was deemed ineligible
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Treatment : Dose Level 6
Number analyzed (Participants) | 38
percentage of patients with response | 89.5 [75.2 to 97.1]

ADVERSE EVENTS:
Time Frame: Baseline to 30 days post treatment, up to 3 years
Description: Some of the observed Adverse Events were collected without regard to the specific Adverse Event Term, but as a general adverse event within an organ system class. These events are noted with the inclusion of "Other, specify" in the term.
Groups:
- Treatment: Trial 1, Dose Level 1: 0.2 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
- Treatment: Trial 1, Dose Level 2: 0.3 mCi/kg Yttrium (Y-90 ibritumomab tiuxetan (IDEC-90Y2B8) IV over 10 minutes on day 8
- Treatment: Trial 2, Dose Level 3; Treatment: Trial 2, Dose Level 4: 50 micrograms/kg Interleukin-11 SC when PLT counts less than 75,000.
- Treatment: Trial 3, Dose Level 5; Treatment: Trial 3, Dose Level 6; Treatment : Phase II (Dose Level 6): 50 micrograms/kg Interleukin-11 SC when PLT counts less than 150,000.
Arm/Group | Treatment: Trial 1, Dose Level 1 | Treatment: Trial 1, Dose Level 2 | Treatment: Trial 2, Dose Level 3 | Treatment: Trial 2, Dose Level 4 | Treatment: Trial 3, Dose Level 5 | Treatment: Trial 3, Dose Level 6 | Treatment : Phase II (Dose Level 6)
Serious Adverse Events (participants affected / at risk) | 4/11 | 5/7 | 4/9 | 2/4 | 1/5 | 1/6 | 6/39
Other Adverse Events (participants affected / at risk) | 11/11 | 7/7 | 9/9 | 4/4 | 5/5 | 6/6 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Trial 1, Dose Level 1 (N=11) | Treatment: Trial 1, Dose Level 2 (N=7) | Treatment: Trial 2, Dose Level 3 (N=9) | Treatment: Trial 2, Dose Level 4 (N=4) | Treatment: Trial 3, Dose Level 5 (N=5) | Treatment: Trial 3, Dose Level 6 (N=6) | Treatment : Phase II (Dose Level 6) (N=39)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (9) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 4 (21) | 2 (6) | 0 (0) | 1 (3) | 1 (3) | 5 (18)
Platelet count decreased (Investigations) | 0 (0) | 2 (12) | 2 (6) | 2 (9) | 0 (0) | 1 (6) | 3 (15)
White blood cell decreased (Investigations) | 0 (0) | 1 (6) | 1 (3) | 0 (0) | 1 (3) | 1 (3) | 3 (12)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Trial 1, Dose Level 1 (N=11) | Treatment: Trial 1, Dose Level 2 (N=7) | Treatment: Trial 2, Dose Level 3 (N=9) | Treatment: Trial 2, Dose Level 4 (N=4) | Treatment: Trial 3, Dose Level 5 (N=5) | Treatment: Trial 3, Dose Level 6 (N=6) | Treatment : Phase II (Dose Level 6) (N=39)
Anemia (Blood and lymphatic system disorders) | 10 (93) | 7 (90) | 9 (57) | 3 (51) | 5 (33) | 6 (72) | 34 (330)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (9) | 0 (0) | 4 (12) | 3 (15) | 4 (12) | 2 (18) | 9 (33)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (15) | 1 (3) | 2 (9) | 1 (3) | 2 (9) | 0 (0) | 5 (18)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (6) | 1 (3) | 2 (9) | 0 (0) | 1 (6) | 0 (0) | 6 (18)
Dry mouth (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (6) | 1 (3) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
Nausea (Gastrointestinal disorders) | 2 (18) | 5 (21) | 3 (9) | 2 (6) | 3 (12) | 2 (6) | 13 (48)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 1 (3) | 2 (6)
Chills (General disorders) | 2 (6) | 0 (0) | 1 (3) | 1 (3) | 1 (6) | 1 (9) | 6 (18)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Fatigue (General disorders) | 2 (9) | 5 (18) | 4 (15) | 1 (3) | 2 (12) | 4 (18) | 21 (84)
Fever (General disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 1 (3) | 1 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (6) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 0 (0) | 2 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 5 (15)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (6) | 1 (3) | 1 (3) | 1 (3) | 2 (6)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (9) | 2 (6) | 6 (21)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Infections and infestations - Other, specify (Infections and infestations) | 6 (18) | 1 (3) | 3 (12) | 0 (0) | 2 (12) | 3 (9) | 11 (36)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Wound infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (6) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Alkaline phosphatase increased (Investigations) | 3 (18) | 1 (6) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 4 (15)
Aspartate aminotransferase increased (Investigations) | 2 (12) | 3 (12) | 1 (6) | 0 (0) | 0 (0) | 2 (9) | 3 (12)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 3 (15)
Cholesterol high (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Neutrophil count decreased (Investigations) | 9 (93) | 6 (141) | 9 (147) | 3 (105) | 5 (60) | 6 (102) | 32 (477)
Platelet count decreased (Investigations) | 10 (129) | 7 (117) | 8 (102) | 4 (84) | 5 (93) | 6 (126) | 39 (711)
Weight gain (Investigations) | 2 (6) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 11 (135) | 7 (192) | 9 (180) | 3 (123) | 5 (72) | 6 (93) | 34 (675)
Anorexia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 5 (21)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (33) | 3 (12) | 4 (30) | 2 (9) | 1 (6) | 5 (18) | 9 (30)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 1 (3) | 1 (6) | 0 (0) | 2 (6) | 5 (15)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (3) | 3 (12) | 1 (6) | 1 (3) | 3 (12) | 10 (33)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 0 (0) | 4 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 3 (18) | 9 (30)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (6) | 2 (6) | 1 (3) | 1 (3) | 1 (3) | 8 (27)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 4 (12)
Depression (Psychiatric disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Gynecomastia (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 2 (6)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (9) | 1 (3) | 0 (0) | 1 (3) | 2 (6) | 3 (9) | 4 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 2 (6) | 2 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 2 (6) | 2 (6) | 0 (0) | 0 (0) | 6 (24)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (3) | 3 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 3 (12) | 2 (6) | 1 (3) | 1 (3) | 5 (15)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (6) | 1 (3) | 1 (3) | 1 (12) | 1 (3) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 2 (9)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hot flashes (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less